CLINICAL TRIAL: NCT02527720
Title: Changing Impulsivity With Mindful Breathing Therapy to Reduce Problem Drinking
Acronym: BBMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Principal Investigator, Carl W. Lejuez, Professor, University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R34AA022213-01A1 (NIH)
Record Dates: First submitted 2015-08-12; First posted 2015-08-19 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Problem Drinking
Keywords: Mindfulness; Therapy; Problem Drinking; Breathing-based mindfulness training
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mindfulness Therapy (Experimental): For the current study the investigators have developed a breathing-based, adapted for feasible application among SUD populations, and easy to carry out in clinical or non-clinical settings referred to as breathing-based mindfulness training (BBMT). BBMT is a simplified form of MM. Its core components are near resonance-frequency breathing (RFB), mindfulness training, positivity and inward attention (more details below).
  Interventions: Behavioral: Mindfulness Therapy

INTERVENTIONS:
Behavioral: Mindfulness Therapy — BBMT is a simplified form of MM. Its core components are near resonance-frequency breathing (RFB), mindfulness training, positivity and inward attention. A key component in BBMT is to be mindful of breathing whenever possible, and breathe at near resonance frequency (RF), known as heart rate variability biofeedback. The human cardiovascular system is known to have resonance characteristics, with the first RF at ~0.1 Hz. RF varies between 4.5 and 7 cycles per minute. Breathing at RF stimulates the cardiovascular system to oscillate at that frequency at a very high amplitude and greatly stimulates the baroreflex system. RFB is known to reduce depression and stress symptoms as well as various diseases related to malfunction of the autonomic nervous system, such as asthma and hypertension.

SUMMARY:
The investigators plan to establish the efficacy of a novel breathing-based mindfulness training (BBMT, a much simplified, easy-to-use version of standard MM) for problem drinking, and test whether impulsivity mediates this effect among a sample of student problem drinkers (i.e., > 8 on AUDIT, the problem drinking Screening Test). The specific aims of this pilot study are as follows:

1. to modify and further develop the easy-to-use BBMT program for directly targeting impulsivity to produce an indirect reduction in problem drinking among college students;
2. to investigate the feasibility and preliminary efficacy of applying BBMT for reducing problem drinking with a pilot randomized controlled trial (RCT);
3. to examine changes in impulsivity, as measured by both behavioral and self-report assessments, as one of the possible mediators in the effect of BBMT on problem drinking, with control for changes in perceived stress and anxiety.

DETAILED DESCRIPTION:
An efficacious strategy for addressing problem substance use among college student drinkers is to target core risk factors. Arguably one of the most clearly documented risk factors for problem drinking among college students is impulsivity, with the relationship holding across various dimensions of impulsivity. Available evidence supports the importance of intervening with impulsivity to limit problem drinking among college students, but there are few proven treatments for any dimension of impulsivity. This notable lack may be due to the traditional view of impulsivity as an unchangeable personality trait. However, recent research suggests personality can change and is sensitive to behavior manipulation. As a result there is clear need for novel approaches targeted at core changes in the individual and their behavior patterns. Mindfulness meditation (MM) is a unique option in this direction as MM is especially useful in reducing impulsive behaviors including problem drinking, but its exact role in affecting different dimensions of impulsivity and in effecting change in problem drinking has yet to be explored. Based on evidence from recent studies, as well as our own pilot work, the investigators hypothesize that one of the mechanisms by which MM reduces problem drinking among college students is by lessening impulsivity - moreover, the focus on changing college student problem drinking is done without any explicit focus on drinking behavior itself. The specific aims of this Stage 1 therapy development study are to: 1) modify and further develop a breathing-based mindfulness therapy (BBMT) for reducing impulsivity and problem drinking among college youth; 2) investigate the feasibility and preliminary efficacy of applying BBMT for reducing problem drinking with a pilot randomized controlled trial (RCT); 3) examine changes in impulsivity, as measured by both behavioral and self-report assessments, as one of possible mediators in the observed effect of BBMT on problem drinking. These aims will be achieved in two phases. In Phase 1 the investigators will expand and fully develop the existing BBMT program with manuals to determine the effective treatment dosage for both problem drinking and impulsivity in an open label trial (n = 10). Using the modified treatment materials from Phase 1, in Phase 2 the investigators will conduct a RCT comparing the effects of modified BBMT to a Supportive Counseling + Progressive Muscle Relaxation (SC + PMR) control condition (n = 36 each) on problem drinking, assessed at baseline, weeks 4 and 8, and a 3-month follow-up. Other potential mediators such as perceived stress and anxiety also will be examined in the final model. This study has great potential implications for reaching college students drinkers less willing to acknowledge their drinking problems as it addresses a core vulnerability (impulsivity) among at-risk students in a manner that limits stigma and may reduce resistance to change. A diverse team experienced in mindfulness, impulsivity and behavior therapy development has been assembled to conduct the proposed R34 project and prepare for a full therapy development study in the future.

ELIGIBILITY:
Inclusion Criteria:

1. UM College Park students aged 18-30
2. AUDIT score of 8 or higher (Babor et al., 2004)
3. A total score on the Barratt Impulsiveness Scale of 73 or higher, which is the mean plus half (1/2) standard deviation, (M=64; SD=17) (Patton et al., 1995)
4. A commitment to adhere to the study protocol with a weekly therapy meeting (about 40 minutes each), and an extra 1.5 to 2 hours for study data collection at week 4 and week 8
5. No plan to move away from the UM campus area for next 2 months

Exclusion Criteria:

1. At current risk of suicide, including suicidal behavior or attempts in the past 30 days
2. A history of schizophrenia or other psychotic disorders
3. Current participation in other clinical studies of addiction or impulsive behavior
4. Severe physical and mental health problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in substance use utilizing the Timeline Follow Back from the baseline to 3 months | Weeks 1-8 and 3 month follow up
  Timeline Follow-back (TLFB) (C. Sobell & B. Sobell, 1992) will be used to record and track participants' recent (past 30 days and 7 days) alcohol-use as well as other drug use frequency. Alcohol-use and other drug use quantity will be recorded for each day on which use was reported. The TLFB method has been shown to have good reliability and validity in college students (Sobell et al., 1989)

SECONDARY OUTCOMES:
Audit | Baseline
  Alcohol Use Diagnostic Identification Test (AUDIT) (Babor et al., 2004), has 10 items which assess frequency of drinking, typical quantity, frequency of heavy drinking, impaired control over drinking, increased salience of drinking, morning drinking, blackouts, and alcohol-related injuries within the past year. A total score of 8 or more has been found to indicate a strong likelihood of hazardous or harmful alcohol consumption
Readiness to Change | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Readiness to Change: Drug and Alcohol version of SOCRATES (Miller & Tonigan, 1996) will be used to evaluate motivation for change
Customary Drinking and Drug Use Record | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Customary Drinking and Drug Use Record (CDDR; Brown et al., 1998) measures lifetime alcohol use and problems to provide a baseline and examine the impact of treatment. The CDDR records age at first use and makes separate lifetime frequency use estimations for beer, wine, and distilled spirits. The CDDR has good reliability for assessing substance use behaviors among adolescents and young adults (Brown et al., 1998) and has been used specifically in college-student samples Doran et al., 2007)
Barratt Impulsiveness Scale | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Barratt Impulsiveness Scale (BIS-11) , includes questions focusing on motor impulsivity (acting without thinking), cognitive impulsivity (making quick cognitive decisions), and future-planning impulsivity (lack of concern about the future), with good internal consistency (alpha = 0.89 to 0.92) and test-retest reliability (0.80). Mean plus one SD in total BIS score from UM study (M = 64; SD = 17) will be used to screen and select those with high impulsivity to be included in this study to assess possible change over time.
UPPS Impulsive Behavioral Scale | Baseline , Week 4 , Week 8, and 3 month Follow Up
  UPPS Impulsive Behavior scale (Whiteside & Lynam, 2001) assesses five personality pathways to impulsive behavior: negative urgency, positive urgency, (lack of) premeditation, (lack of) perseverance, and sensation seeking
Delay Discounting of Hypothetical Money Gains | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Delay Discounting of Hypothetical Money Gains, is a computerized binary-choice procedure. On each trial, two outcomes will be presented on the screen: one is an amount of money available immediately; the other is a larger amount of money ($50, $1,000) available after some delay (1 week, 1 year, etc.). The computerized algorithm (Holt et al., 2003) will adjust the immediate outcome for each amount/delay pairing over 6 trials to determine an indifference point, resulting in 6 indifference points (corresponding to the 6 delays) for each of 2 amounts ($50, $1,000).
Stop-Signal Task (SST) | Baseline , Week 4 , Week 8, and 3 month Follow Up
  A personal computer will be used to conduct the SST, which presents two types of trials: GO and STOP. In GO trials, participants will respond with a keystroke as quickly as possible following the presentation of a visual go stimulus. In STOP trials (25% of all trials), an auditory stop signal will follow the presentation of the visual go signal. Subjects will be instructed to inhibit the go response on hearing the stop signal. The latency between onset of the go and stop signals will be titrated in the following manner: failure on a STOP trial will result in a 50ms increase in this latency, and success will result in a 50ms decrease. This method will converge on a latency, the stop signal delay (SSD) at which a participant succeeds on half of all STOP trials. After 16 GO practice trials, participants will complete five blocks of 64 trials.
Spielberger State-Trait Anxiety Inventory (STAI): | Baseline , Week 4 , Week 8, and 3 month Follow Up
  both trait and state anxiety will be measured monthly to monitor changes over time
The Center for Epidemiological Studies Depression Scale (CES-D) | Baseline , Week 4 , Week 8, and 3 month Follow Up
  The Center for Epidemiological Studies Depression Scale (CES-D) (Radloff, 1977) is a 20-item self-report inventory measuring mood and symptoms of depression.
Perceived Stress Scale | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Perceived Stress Scale is a global measure of perceived stress in daily life (Chiang et al., 2005) designed to gauge the degree to which common situations are appraised as stressful
Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) is a well-validated 36-item, self-report questionnaire that assesses multiple aspects of emotion dysregulation. The DERS yields a total score that is comprised of scores on six subscales: nonacceptance of emotional responses, lack of emotional awareness, impulse control difficulties, difficulties engaging in goal directed behavior, lack of emotional clarity, and limited access to emotion regulation strategies.
Five-Facet Mindfulness Questionnaire | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Five-Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2006) is an instrument based on factor analysis of five independently developed mindfulness scales. The five factors appear to represent elements of mindfulness as it is currently conceptualized. The five facets are observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. The FFMQ is one of the most popular scales used in study of mindfulness.
Perceived Quality of Life Measure | Baseline , Week 4 , Week 8, and 3 month Follow Up
  Perceived Quality of Life Measure (Burckhardt & Anderson, 2003) will be employed to assess general well-being. These measures will be given at baseline and every 4 weeks during treatment.
Therapist adherence and competence | Week 4, Week 8, and 3 month Follow Up
  Therapist adherence and competence. During the open trial all treatment sessions will be audio taped and rated by independent raters (e.g., not associated with treatment delivery) so as to assess therapist adherence to the treatment protocol. Specific therapist behaviors will be considered "prescribed" and "proscribed" (Waltz et al., 1993) in order to assure that BBMT and SC + PMR treatment are distinct. Drs. Chen and Lejuez will review 20% of the audiotapes to maintain reliability. If therapist drift from the protocol is detected, the problem will be discussed in staff meetings and corrected through supervision.
The Program Evaluation Form | Week 4, Week 8, and 3 month Follow Up
  he Program Evaluation Form is an 8-item self-report measure assessing participants' perceptions of and satisfaction with the treatment services.
Working Alliance Inventory (WAI) | Week 4, Week 8
  he Working Alliance Inventory (WAI) (Horvath & Greenberg, 1989) will be used to assess therapeutic alliance. The WAI is a 36-item measure composed of items reflecting desirable aspects of the therapeutic relationship. Each item is assessed on a 7-point Likert scale ranging from 1 (never) to 7 (always), with higher scores indicating more positive therapeutic alliance.
RFB or MM Feedback and Quality Assessment | Weeks 1-8 and 3 month follow up
  RFB or MM Feedback and Quality Assessment: BBMT participants will report daily quantity and quality of RFB or MM practice
Treatment Progress/Completion | Week 8
  Treatment Progress/Completion: A checklist for the therapist to document the proportion of training components being delivered and practiced by the end of week 8 facilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Lejuez, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- 2103 Cole Field House, College Park, Maryland, United States

REFERENCES:
- [Background] Chen KW, Comerford A, Shinnick P, Ziedonis DM. Introducing qigong meditation into residential addiction treatment: a pilot study where gender makes a difference. J Altern Complement Med. 2010 Aug;16(8):875-82. doi: 10.1089/acm.2009.0443. PMID 20649456
- [Background] Carroll, K. M., & Nuro, K. F. (2002). One size cannot fit all: A stage model for psychotherapy manual development. Clinical Psychology: Science and Practice, 9(4), 396-406.
- [Background] Karavidas MK, Lehrer PM, Vaschillo E, Vaschillo B, Marin H, Buyske S, Malinovsky I, Radvanski D, Hassett A. Preliminary results of an open label study of heart rate variability biofeedback for the treatment of major depression. Appl Psychophysiol Biofeedback. 2007 Mar;32(1):19-30. doi: 10.1007/s10484-006-9029-z. Epub 2007 Mar 1. PMID 17333315
- [Background] Lehrer PM, Vaschillo E, Vaschillo B. Resonant frequency biofeedback training to increase cardiac variability: rationale and manual for training. Appl Psychophysiol Biofeedback. 2000 Sep;25(3):177-91. doi: 10.1023/a:1009554825745. PMID 10999236
- [Background] Schein MH, Gavish B, Herz M, Rosner-Kahana D, Naveh P, Knishkowy B, Zlotnikov E, Ben-Zvi N, Melmed RN. Treating hypertension with a device that slows and regularises breathing: a randomised, double-blind controlled study. J Hum Hypertens. 2001 Apr;15(4):271-8. doi: 10.1038/sj.jhh.1001148. PMID 11319676
- [Background] Krueger, R. A. (1994). Focus groups: A practical guide for applied research. Sage
- [Background] Krueger, R. A., & Casey, M. A. (2009). Focus groups: A practical guide for applied research (2 e.d.). Sage.
- [Background] Strauss, A., & Corbin, J. M. (1997). Grounded theory in practice. Sage.